CLINICAL TRIAL: NCT01809964
Title: Clinical Trial to Evaluate ANT-1401 in Subjects With Lateral Canthal Lines
Brief Title: Clinical Trial to Evaluate ANT-1401 in Crow's Feet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterios Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANT-1401-LCL-203
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-12

CONDITIONS: Lateral Canthal Lines; Crows Feet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental): ANT-1401
  Interventions: Biological: ANT-1401
- Dose 2 (Experimental): ANT-1401
  Interventions: Biological: ANT-1401
- Vehicle (Placebo Comparator): Placebo Vehicle
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: ANT-1401
  Arms: Dose 1; Dose 2
Biological: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to confirm the effect of ANT-1401 in the treatment of Lateral Canthal Lines.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 60 years of age
* mild to moderate Crow's Feet wrinkles (IGA 1-2) at rest
* moderate to severe Crow's Feet (IGA 2-3) on contraction
* moderate to severe Crow's Feet (SSA 2-3) on contraction
* Have adequate vision to assess facial wrinkles in a mirror

Exclusion Criteria:

* botulinum toxin treatment in the prior 6 months
* history of periocular surgery, brow lift or related procedures
* soft tissue augmentation in the lateral canthal region in the prior 12 months
* dermabrasion or laser treatment in the periocular region in the last 6 months
* topical prescription-strength retinoids in the prior 3 months
* present or history of neuromuscular disease
* present or history of "dry eye"
* systemic aminoglycoside use in the week prior to treatment application

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment Scale | Week 4

SECONDARY OUTCOMES:
Subject Self-Assessment | Week 4

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Birmingham, Alabama
  - Miami, Florida
  - Pinellas Park, Florida
  - West Palm Beach, Florida
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Knoxville, Tennessee